CLINICAL TRIAL: NCT00698828
Title: A Phase 2b, Multicenter, Randomized, Double-Blind, Parallel, Placebo-Controlled Study to Evaluate the Efficacy and Safety of SUN11031 for Injection Administered Subcutaneously Twice Daily for 12 Weeks to Subjects Having Cachexia Associated With Chronic Obstructive Pulmonary Disease
Brief Title: SUN11031 in Cachexia Associated With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASBI 307
Record Dates: First submitted 2008-05-01; First posted 2008-06-17 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Cachexia
Keywords: Cachexia, COPD, Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Cachexia; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): SUN11031 for injection, low dose, twice daily for 12 weeks
  Interventions: Drug: SUN11031 20 μg/kg
- Group 2 (Experimental): SUN11031 for injection, higher dose, twice daily for 12 weeks
  Interventions: Drug: SUN11031 40 μg/kg
- Group 3 (Placebo Comparator): Placebo injection, twice daily for 12 weeks
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Placebo comparator — Twice daily subcutaneous injections of placebo for 12 weeks.
  Arms: Group 3
Drug: SUN11031 20 μg/kg — Twice daily subcutaneous injections of SUN11031 20 μg/kg for 12 weeks.
  Arms: Group 1
Drug: SUN11031 40 μg/kg — Twice daily subcutaneous injections of SUN11031 40 μg/kg for 12 weeks.
  Arms: Group 2

SUMMARY:
To evaluate SUN11031 for subcutaneous injection compared to placebo in subjects with cachexia associated with Chronic Obstructive Pulmonary Disease (COPD) to determine the effect on physical performance and body composition.

ELIGIBILITY:
Inclusion Criteria:

Each participant had to meet the following criteria to be enrolled in the study:

1. Male or non-pregnant female participants 50 years or older with a clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD) for greater than or equal to 12 months
2. Walked a distance of greater than or equal to 100 but less than or equal to 450 meters during the 6-Minute Walk Test (MWT) performed at screening.
3. Chest x-ray within the past year that was compatible with COPD
4. Documented involuntary nonedematous weight loss of greater than 5% of participant's usual body weight over the past 12 months or BMI less than or equal to 21 kg/m^2 for males or Body Mass Index (BMI) less than or equal to 20 kg/m^2 for females
5. Female participants who were clinically sterile (eg, either postmenopausal or had undergone a tubal ligation or hysterectomy) or were practicing a medically acceptable method of birth control (eg, oral, transdermal, implantable, or injectable contraceptive medications; double-barrier method or intrauterine device)

Exclusion Criteria:

Participants who met any of the following criteria were excluded from the study:

1. BMI greater than 26 kg/m^2
2. Used, over a total of 7 or more days, parenteral corticosteroids at a dose equivalent to prednisone at greater than or equal to 5 mg/day or oral corticosteroids at a dose equivalent to prednisone at greater than 10 mg/day within the 2 months before screening; however, participants were allowed to participate if on stable doses equivalent to prednisone at less than or equal to 10 mg/day for at least 2 months before screening, and were planning to remain on the same stable dose throughout the study
3. Were planning to start a pulmonary rehabilitation program during the study (participant may have been enrolled in the study if he or she was currently on a stable maintenance program)
4. Weight loss that was considered to be, in the opinion of the investigator, the result of food deprivation
5. Unintended weight loss that may have been due to disease other than COPD
6. Unable or unwilling to be trained to self-administer the study drug by subcutaneous injection bid, and for whom arrangements could not be made for a third party to reliably administer the injections
7. Severe anemia (hemoglobin less than or equal to 8 g/dL)
8. COPD exacerbation defined as a Type 1 or 2 exacerbation according to the Winnipeg criteria, acute infection, or prolonged fever within 4 weeks before screening
9. Undergoing treatment or evaluation for cancer, or had a history of treatment for cancer within the past 3 years, exception being nonmelanoma skin cancer (basal cell or squamous cell carcinoma of the skin) and carcinoma in situ of the cervix
10. Type I or type II diabetes mellitus or a fasting serum glucose of greater than or equal to 115 mg/dL (6.4 mmol/L) (fasting was overnight)
11. Serious disease or conditions that would have interfered with the participant's ability to complete the functional measures included in this protocol; or any illness that, in the opinion of the investigator, might have interfered with the results of the study or the participant's ability to participate
12. Pulmonary embolism, deep venous thrombosis, or clinically significant primary pulmonary hypertension within the past 6 months
13. Significant ischemic heart disease or chronic heart failure (New York Heart Association Class IV cardiac disease)
14. Uncontrolled hypertension (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 110 mm Hg)
15. A history of symptomatic orthostatic hypotension or syncope; or orthostatic hypotension at screening or baseline (Days -6 to -3) (orthostatic hypotension was defined as a decrease in systolic blood pressure by greater than or equal to 20 mm Hg measured after 2 minutes in a standing position compared with the systolic blood pressure measured after 10 minutes in a supine position)
16. Evidence of ascites, pleural effusion, or lower extremity edema
17. Severe vitamin D deficiency (25-hydroxyvitamin D less than 10 ng/mL)
18. Known mechanical obstruction of the alimentary tract and/or malabsorption
19. Dental or swallowing problems that may have had a negative effect on food intake
20. Serum creatinine greater than 2.5 mg/dL; or alanine aminotransferase, aspartate aminotransferase, or gamma-glutamyl transferase greater than 3 times the upper limit of normal, or bilirubin greater than 2.5 mg/dL
21. A diagnosis of human immunodeficiency virus infection or AIDS
22. Used any prescription drugs and non-prescription drugs/herbs that cause weight loss or affect appetite and absorption or that may cause nausea; or used appetite-promoting or anabolic medications within 15 days before screening
23. A history of alcohol or drug abuse that, in the opinion of the investigator, would have interfered with the participant's ability to comply with the dosing schedule and protocol-specified requirements
24. Hypersensitive to any component of SUN11031, or participated at any time in any study in which SUN11031 was administered
25. Received an investigational drug or product, or participated in a drug study within 30 days before screening
26. Non-ambulatory or unwilling to cooperate fully with the investigator or a designee, or unwilling or unable to comply with study requirements, such as all assessments required by the protocol, including completion of measures for functional capacity and pulmonary function, or frequent blood sampling and meal instructions; or unable or unwilling to attend all study visits

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2008-05-15 (Actual); Primary Completion 2009-10-08 (Actual); Study Completion 2009-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (43):
- United States (11):
  - Waterbury Pulmonary Associates, Waterbury, Connecticut
  - Clinical Research of West Florida, Clearwater, Florida
  - Innovative Research of West Florida, Largo, Florida
  - The Center for Clinical Research, Washington County Hospital, Hagerstown, Maryland
  - Montana Medical Research, Inc., Missoula, Montana
  - The Asthma & Allergy Center, Papillion, Nebraska
  - Health Science Research Center - Asthma & Allergy Associates, Cortland, New York
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Pulmonary Consultants, Tacoma, Washington
- Argentina (18):
  - Centro de Investigaciones Médicas, Florencío Varela, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata, Buenos Aires
  - Centro Respiratorio Quilmes, Quilmes, Buenos Aires
  - Instituto de Investigaciones Clínicas Cipolletti, Cipolletti, Río Negro Province
  - Clinica del Tórax, Rosario, Santa Fe Province
  - Instituto Cardiovascular de Rosario, Rosario, Santa Fe Province
  - CEMIT, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigación Médica Lanús, Buenos Aires
  - FAICEP, Capital Federal
  - Instituto Médico de Asistencia e Investigación, Capital Federal
  - Centro Médico Dra. De Salvo, Capital Federal
  - Centro Médico Belgrano, Capital Federal
  - Centro Ceri, Capital Federal
  - Centro de Estudios Neumonologicos, Capital Federal
  - Fuesmen, Mendoza
  - Instituto de Enfermedades Respiratorias, Mendoza
  - Centro de Medicina Respiratoria, Paraná
  - Instituto de Patologia Respiratoria, San Miguel de Tucumán
- Chile (3):
  - Hospital Barros Luco Trudeau, Santiago
  - Hospital San Jose, Santiago
  - Integramedica La Florida, Santiago
- Guatemala (4):
  - Instituto Pneos, Guatemala City
  - Edificio Centro Medico II, Guatemala City
  - Private Clinic, Guatemala City
  - Edificio Medico San Lucas, Quetzaltenango
- Honduras (2):
  - Centro de Neumologia y Alergia, San Pedro Sula
  - Instituto Nacional Cardiopulmonar, Tegucigalpa
- Romania (5):
  - Spitalul Clinic de Pneumoftiziologie "Leon Daniello" Cluj-Napoca, Cluj-Napoca, Cluj
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologoe "Dr. Victor Babes", Timișoara, Timiș County
  - Spitalul Clinic de Pneumoftiziologie "Leon Daniello" Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic de Pneumoftiziologie Constanta, Cartier Palazul Mare, Constanța
  - Spitalul Clinic Judetean Sibiu, Clinica Medicala, Sibiu

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- See also: Related Info — http://www.nhlbi.nih.gov/health/dci/Diseases/Copd/Copd_WhatIs.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 227 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 11 clinic sites in the United States of America (USA), 19 in Argentina, 3 in Chile, 4 in Guatemala, 2 in Honduras, and 6 in Romania. Three (3) participants were enrolled but not treated with the study drug. The remaining 224 enrolled participants were teated.
Pre-assignment Details: Spirometry was performed on participants during screening to define the pulmonary function of each participating subject enrolled in this study.
Groups:
- Placebo: Participants with chronic obstructive pulmonary disease who were administered SUN11031-matching placebo subcutaneous injections twice daily for 12 weeks.
- SUN11031 20 μg/kg: Participants with chronic obstructive pulmonary disease who were administered SUN11031 20 μg/kg subcutaneous injections twice daily for 12 weeks.
- SUN11031 40 μg/kg: Participants with chronic obstructive pulmonary disease who were administered SUN11031 40 μg/kg subcutaneous injections twice daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg
Started | 76 | 75 | 76
Completed | 67 | 60 | 65
Not Completed | 9 | 15 | 11
Not completed — Adverse Event | 3 | 4 | 4
Not completed — Death | 0 | 0 | 1
Not completed — Exacerbation of COPD | 1 | 3 | 0
Not completed — Exacerbation of COPD (Not treated) | 1 | 0 | 0
Not completed — Investigator/Sponsor decision | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrew consent | 0 | 7 | 4
Not completed — Withdrew consent (not treated) | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg | Total
Number analyzed (Participants) | 73 | 75 | 76 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (8.85) | 64.5 (8.03) | 66.2 (9.20) | 65.6 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 24 | 24 | 79
  Male | 42 | 51 | 52 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 63 | 59 | 179
  Not Hispanic or Latino | 16 | 12 | 17 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 65 | 67 | 71 | 203
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Day 85 in the Distance Walked During the 6 Minute Walk Test (MWT) Following Treatment With SUN11031 in Participants Having Cachexia Associated With Chronic Obstructive Pulmonary Disease (COPD)
Description: Assessment of functional capacity in study participants with chronic obstructive pulmonary disease (COPD) via the 6-minute walk test (6MWT) provided an objective measure of disability. The 6MWT is a practical and objective evaluation of functional exercise capacity. The test measures the distance that a participant can quickly walk on a flat, hard surface in 6 minutes. In order to ensure uniformity among the sites, the specifications of the course for the 6MWT were modified from being 30 meters long with 60-meter laps to be 15 meters long with 30-meter laps to accommodate space limitations encountered at select sites.
Time Frame: Baseline up to Day 85 post dose.
Population: Distance walked during the 6 Minute Walk Test was assessed using the Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg
Number analyzed (Participants) | 72 | 73 | 69
meters
  Baseline | 317.30 (80.62) | 333.93 (78.91) | 333.30 (68.20)
  Change at Day 85 | 28.50 (54.72) | 5.85 (53.38) | 10.04 (62.16)

2. Secondary Outcome: Mean Change From Baseline to Days 29, 57, and 85 in the Distance Walked During the 6 Minute Walk Test (MWT) Following Treatment With SUN11031 in Participants Having Cachexia Associated With Chronic Obstructive Pulmonary Disease (COPD)
Description: as for outcome 1
Time Frame: Baseline up to Day 29, Day 57, and Day 85 post dose.
Population: Distance walked during the 6 Minute Walk Test was assessed using the Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg
Number analyzed (Participants) | 72 | 73 | 69
meters
  Baseline | 317.30 (80.62) | 333.93 (78.91) | 333.30 (68.20)
  Change at Day 29 | 24.26 (56.41) | 2.80 (46.45) | 15.40 (44.39)
  Change at Day 57 | 27.80 (50.46) | 9.66 (47.80) | 17.46 (48.27)
  Change at Day 85 | 28.50 (54.72) | 5.85 (53.38) | 10.04 (62.16)

3. Secondary Outcome: Mean Change From Baseline to Days 29, 57, and 85 in the Distance Walked During the 6 Minute Walk Test (MWT) By Sub-groups Following Treatment With SUN11031 in Participants Having Cachexia Associated With Chronic Obstructive Pulmonary Disease (COPD)
Description: as for outcome 1
Time Frame: Baseline up to Day 29, Day 57, and Day 85 post dose.
Population: Distance walked during the 6 Minute Walk Test was assessed using the Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg
Number analyzed (Participants) | 72 | 73 | 69
meters
  Males: Baseline: number analyzed (Participants) | 41 | 51 | 48
  Males: Baseline | 316.07 (78.64) | 336.24 (86.36) | 337.95 (64.10)
  Males: Change at Day 29: number analyzed (Participants) | 41 | 51 | 48
  Males: Change at Day 29 | 30.06 (50.34) | -0.97 (53.57) | 11.56 (44.91)
  Males: Change at Day 57: number analyzed (Participants) | 41 | 51 | 48
  Males: Change at Day 57 | 30.41 (38.30) | 10.08 (54.74) | 11.13 (45.14)
  Males: Change at Day 85: number analyzed (Participants) | 41 | 51 | 48
  Males: Change at Day 85 | 33.24 (49.15) | 4.17 (61.90) | 11.05 (46.17)
  Females: Baseline: number analyzed (Participants) | 31 | 22 | 21
  Females: Baseline | 318.94 (84.44) | 328.60 (59.58) | 322.67 (77.39)
  Females: Change at Day 29: number analyzed (Participants) | 31 | 22 | 21
  Females: Change at Day 29 | 16.53 (63.69) | 11.55 (21.19) | 24.42 (42.91)
  Females: Change at Day 57: number analyzed (Participants) | 31 | 22 | 21
  Females: Change at Day 57 | 24.34 (63.63) | 8.70 (26.45) | 31.94 (53.09)
  Females: Change at Day 85: number analyzed (Participants) | 31 | 22 | 21
  Females: Change at Day 85 | 22.23 (61.60) | 9.75 (25.06) | 7.75 (90.11)
  Younger Than 65 years: Baseline: number analyzed (Participants) | 30 | 36 | 30
  Younger Than 65 years: Baseline | 353.89 (78.95) | 353.35 (72.62) | 353.30 (70.19)
  Younger Than 65 years: Change at Day 29: number analyzed (Participants) | 30 | 36 | 30
  Younger Than 65 years: Change at Day 29 | 33.30 (73.90) | 5.19 (43.01) | 28.31 (48.78)
  Younger Than 65 years: Change at Day 57: number analyzed (Participants) | 30 | 36 | 30
  Younger Than 65 years: Change at Day 57 | 36.50 (60.86) | 11.79 (47.78) | 24.38 (62.35)
  Younger Than 65 years: Change at Day 85: number analyzed (Participants) | 30 | 36 | 30
  Younger Than 65 years: Change at Day 85 | 31.29 (66.54) | 8.76 (46.19) | 9.13 (81.60)
  65 Years and older: Baseline: number analyzed (Participants) | 42 | 37 | 39
  65 Years and older: Baseline | 291.17 (71.88) | 315.04 (81.14) | 317.92 (63.29)
  65 Years and older: Change at Day 29: number analyzed (Participants) | 42 | 37 | 39
  65 Years and older: Change at Day 29 | 17.87 (39.56) | 0.47 (50.05) | 4.92 (38.00)
  65 Years and older: Change at Day 57: number analyzed (Participants) | 42 | 37 | 39
  65 Years and older: Change at Day 57 | 21.58 (41.16) | 7.59 (48.39) | 12.14 (33.71)
  65 Years and older: Change at Day 85: number analyzed (Participants) | 42 | 37 | 39
  65 Years and older: Change at Day 85 | 26.51 (45.22) | 3.02 (60.08) | 10.75 (42.79)
  Body Mass Index (BMI) <18.9 kg/m^2: Baseline: number analyzed (Participants) | 40 | 36 | 27
  Body Mass Index (BMI) <18.9 kg/m^2: Baseline | 313.28 (83.74) | 322.42 (85.37) | 328.58 (74.00)
  Body Mass Index (BMI) <18.9 kg/m^2: Change at Day 29: number analyzed (Participants) | 40 | 36 | 27
  Body Mass Index (BMI) <18.9 kg/m^2: Change at Day 29 | 15.78 (45.55) | 6.46 (41.74) | 16.31 (54.65)
  Body Mass Index (BMI) <18.9 kg/m^2: Change at Day 57: number analyzed (Participants) | 40 | 36 | 27
  Body Mass Index (BMI) <18.9 kg/m^2: Change at Day 57 | 17.06 (51.79) | 9.67 (47.08) | 12.37 (54.52)
  Body Mass Index (BMI) <18.9 kg/m^2: Change at Day 85: number analyzed (Participants) | 40 | 36 | 27
  Body Mass Index (BMI) <18.9 kg/m^2: Change at Day 85 | 14.51 (55.14) | 5.21 (54.06) | 24.99 (48.12)
  Body Mass Index (BMI) ≥18.9 kg/m^2: Baseline: number analyzed (Participants) | 32 | 37 | 42
  Body Mass Index (BMI) ≥18.9 kg/m^2: Baseline | 322.33 (77.56) | 345.14 (71.47) | 336.34 (64.94)
  Body Mass Index (BMI) ≥18.9 kg/m^2: Change at Day 29: number analyzed (Participants) | 32 | 37 | 42
  Body Mass Index (BMI) ≥18.9 kg/m^2: Change at Day 29 | 34.93 (66.93) | -0.76 (50.94) | 14.81 (37.21)
  Body Mass Index (BMI) ≥18.9 kg/m^2: Change at Day 57: number analyzed (Participants) | 32 | 37 | 42
  Body Mass Index (BMI) ≥18.9 kg/m^2: Change at Day 57 | 41.22 (46.08) | 9.65 (49.15) | 20.74 (44.18)
  Body Mass Index (BMI) ≥18.9 kg/m^2: Change at Day 85: number analyzed (Participants) | 32 | 37 | 42
  Body Mass Index (BMI) ≥18.9 kg/m^2: Change at Day 85 | 45.99 (49.65) | 6.47 (53.47) | 0.44 (68.54)
  Forced Expiratory Volume in 1 second (FEV1) <37% predicted: Baseline: number analyzed (Participants) | 38 | 40 | 28
  Forced Expiratory Volume in 1 second (FEV1) <37% predicted: Baseline | 296.61 (82.27) | 315.35 (89.66) | 320.20 (75.06)
  Forced Expiratory Volume in 1 second (FEV1) <37% predicted: Cange at Day 29: number analyzed (Participants) | 38 | 40 | 28
  Forced Expiratory Volume in 1 second (FEV1) <37% predicted: Cange at Day 29 | 28.65 (48.12) | -8.20 (52.10) | 16.31 (39.96)
  Forced Expiratory Volume in 1 second (FEV1) <37% predicted: Change at Day 57: number analyzed (Participants) | 38 | 40 | 28
  Forced Expiratory Volume in 1 second (FEV1) <37% predicted: Change at Day 57 | 27.67 (49.80) | 1.94 (54.31) | 15.52 (47.63)
  Forced Expiratory Volume in 1 second (FEV1) <37% predicted: Change at Day 85: number analyzed (Participants) | 38 | 40 | 28
  Forced Expiratory Volume in 1 second (FEV1) <37% predicted: Change at Day 85 | 20.87 (51.34) | -6.17 (58.31) | 2.23 (80.61)
  Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted: Baseline: number analyzed (Participants) | 34 | 33 | 41
  Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted: Baseline | 340.43 (73.14) | 356.46 (57.08) | 342.25 (62.47)
  Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted: Change at Day 29: number analyzed (Participants) | 34 | 33 | 41
  Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted: Change at Day 29 | 19.61 (64.46) | 16.13 (34.82) | 14.82 (47.47)
  Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted: Change at Day 57: number analyzed (Participants) | 34 | 33 | 41
  Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted: Change at Day 57 | 27.93 (51.94) | 19.02 (37.19) | 18.79 (49.25)
  Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted: Change at Day 85: number analyzed (Participants) | 34 | 33 | 41
  Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted: Change at Day 85 | 37.02 (57.85) | 20.42 (43.24) | 15.38 (45.94)

4. Secondary Outcome: Number of Participants With Improvement in Distance Walked During the 6 Minute Walk Test (MWT) By Sub-groups Following Treatment With SUN11031 in Participants Having Cachexia Associated With Chronic Obstructive Pulmonary Disease
Description: as for outcome 1
Time Frame: Baseline up to Day 85 post dose.
Population: The number of participants with improved walking distance was assessed using the Intent-to-Treat population.
Measure: Number; unit: participants
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg
Number analyzed (Participants) | 72 | 73 | 69
participants
  ≥20 meter improvement at Day 85 : Males: number analyzed (Participants) | 41 | 51 | 48
  ≥20 meter improvement at Day 85 : Males | 21 | 30 | 22
  ≥20 meter improvement at Day 85 : Females: number analyzed (Participants) | 31 | 22 | 21
  ≥20 meter improvement at Day 85 : Females | 17 | 6 | 12
  ≥20 meter improvement at Day 85 : Younger than 65 years: number analyzed (Participants) | 30 | 36 | 30
  ≥20 meter improvement at Day 85 : Younger than 65 years | 15 | 13 | 15
  ≥20 meter improvement at Day 85 : 65 Years and older: number analyzed (Participants) | 42 | 37 | 39
  ≥20 meter improvement at Day 85 : 65 Years and older | 23 | 13 | 19
  ≥20 meter improvement at Day 85 : BMI <18.9 kg/m^2: number analyzed (Participants) | 40 | 36 | 27
  ≥20 meter improvement at Day 85 : BMI <18.9 kg/m^2 | 17 | 12 | 18
  ≥20 meter improvement at Day 85 : BMI ≥18.9 kg/m^2: number analyzed (Participants) | 32 | 37 | 42
  ≥20 meter improvement at Day 85 : BMI ≥18.9 kg/m^2 | 21 | 14 | 16
  ≥20 meter improvement at Day 85 : Forced Expiratory Volume in 1 second (FEV1) <37% predicted: number analyzed (Participants) | 38 | 40 | 28
  ≥20 meter improvement at Day 85 : Forced Expiratory Volume in 1 second (FEV1) <37% predicted | 16 | 11 | 14
  ≥20 meter improvement at Day 85 : Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted: number analyzed (Participants) | 34 | 33 | 41
  ≥20 meter improvement at Day 85 : Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted | 22 | 15 | 20
  ≥10 meter improvement at Day 85 : Males: number analyzed (Participants) | 41 | 51 | 48
  ≥10 meter improvement at Day 85 : Males | 28 | 24 | 26
  ≥10 meter improvement at Day 85 : Females: number analyzed (Participants) | 31 | 22 | 21
  ≥10 meter improvement at Day 85 : Females | 22 | 10 | 14
  ≥10 meter improvement at Day 85 : Younger than 65 years: number analyzed (Participants) | 30 | 36 | 30
  ≥10 meter improvement at Day 85 : Younger than 65 years | 20 | 17 | 19
  ≥10 meter improvement at Day 85 : 65 Years and older: number analyzed (Participants) | 42 | 37 | 39
  ≥10 meter improvement at Day 85 : 65 Years and older | 30 | 17 | 21
  ≥10 meter improvement at Day 85 : BMI <18.9 kg/m^2: number analyzed (Participants) | 40 | 36 | 27
  ≥10 meter improvement at Day 85 : BMI <18.9 kg/m^2 | 24 | 16 | 19
  ≥10 meter improvement at Day 85 : BMI ≥18.9 kg/m^2: number analyzed (Participants) | 32 | 37 | 42
  ≥10 meter improvement at Day 85 : BMI ≥18.9 kg/m^2 | 26 | 18 | 21
  ≥10 meter improvement at Day 85 : Forced Expiratory Volume in 1 second (FEV1) <37% predicted: number analyzed (Participants) | 38 | 40 | 28
  ≥10 meter improvement at Day 85 : Forced Expiratory Volume in 1 second (FEV1) <37% predicted | 24 | 16 | 15
  ≥10 meter improvement at Day 85 : Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted: number analyzed (Participants) | 34 | 33 | 41
  ≥10 meter improvement at Day 85 : Forced Expiratory Volume in 1 second (FEV1) ≥37% predicted | 26 | 18 | 25

5. Secondary Outcome: Mean Change in Body Weight From Baseline Through Day 99 Following Treatment With SUN11031 in Participants Having Cachexia Associated With Chronic Obstructive Pulmonary Disease
Description: Measurements of body weight were performed in the morning when the participant had an empty stomach (ie, had consumed no food overnight) and had emptied the bladder and had a bowel movement, if possible. These measurements were performed using the same calibrated scale for an individual participant throughout study.
Time Frame: Baseline up to Day 8, Day 15, Day 22, Day 29, Day 43, Day 57, Day 85, and Day 99 post dose.
Population: Mean change in body weight was assessed using the Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg
Number analyzed (Participants) | 72 | 73 | 69
kg
  Baseline | 48.93 (7.89) | 50.63 (8.69) | 53.16 (8.80)
  Change at Day 8 | 0.31 (0.72) | 0.78 (0.77) | 1.00 (0.90)
  Change at Day 15 | 0.43 (0.93) | 1.09 (1.28) | 1.34 (1.12)
  Change at Day 22 | 0.44 (1.14) | 1.36 (1.40) | 1.68 (1.42)
  Change at Day 29 | 0.53 (1.23) | 1.43 (1.56) | 1.86 (1.51)
  Change at Day 43 | 0.48 (1.42) | 1.62 (1.68) | 2.03 (1.63)
  Change at Day 57 | 0.66 (1.47) | 1.62 (1.81) | 2.15 (1.86)
  Change at Day 85 | 0.90 (1.71) | 1.75 (2.27) | 2.44 (2.18)
  Change at Day 99 | 0.84 (1.72) | 1.38 (2.35) | 1.88 (1.96)

6. Secondary Outcome: Mean Change in Lean Body Mass From Baseline Through Days 29, 85 and 99 Following Treatment With SUN11031 in Participants Having Cachexia Associated With Chronic Obstructive Pulmonary Disease
Description: Lean body mass was assessed based on whole-body dual-energy x-ray absorptiometry (DXA).
Time Frame: Baseline up to Day 29, Day 85, and Day 99 post dose.
Population: Mean change in lean body mass was assessed using the Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg
Number analyzed (Participants) | 72 | 73 | 69
kg
  Baseline | 37.85 (6.77) | 39.25 (7.75) | 40.39 (6.80)
  Change at Day 29 | 0.45 (0.95) | 1.12 (1.13) | 1.32 (1.01)
  Change at Day 85 | 0.29 (1.06) | 1.36 (1.24) | 1.44 (1.50)
  Change at Day 99 | 0.22 (1.16) | 0.90 (1.27) | 0.74 (1.55)

7. Secondary Outcome: Absolute Concentrations of SUN11031 Following Treatment With SUN11031 in Participants Having Cachexia Associated With Chronic Obstructive Pulmonary Disease
Description: Absolute concentrations of SUN11031 in participant plasma samples were measured. When participants were randomly assigned into 1 of 3 treatment groups at baseline, they were also randomly assigned into 1 of 2 sequences in the pharmacokinetic (PK) sparse sampling schedule based on the randomization number.
Time Frame: Day 1 and Day 85 pre-dose; Day 1 at 1 hour and 4 hours; Day 29 at 0.08 hours and 1.5 hours; Day 57 at 0.08 hours and 6 hours; Day 85 at 0.5 hours and 3 hours postdose.
Population: Absolute concentrations of SUN11031 were assessed using the pharmacokinetic population.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg
Number analyzed (Participants) | 73 | 74 | 76
pg/mL
  Seq 1: Predose 0 hrs, Day 1: number analyzed (Participants) | 35 | 35 | 32
  Seq 1: Predose 0 hrs, Day 1 | 49.09 (41.92) | 392.00 (2032.51) | 2125.02 (9355.92)
  Seq 2: Predose 0 hrs, Day 1: number analyzed (Participants) | 35 | 33 | 38
  Seq 2: Predose 0 hrs, Day 1 | 58.93 (94.06) | 1083.62 (5600.63) | 79.49 (105.07)
  Seq 1+2: Predose 0 hrs, Day 1: number analyzed (Participants) | 70 | 68 | 70
  Seq 1+2: Predose 0 hrs, Day 1 | 54.01 (72.46) | 727.64 (4147.16) | 1014.59 (6354.99)
  Seq 1: Predose 0 hrs, Day 85: number analyzed (Participants) | 31 | 28 | 29
  Seq 1: Predose 0 hrs, Day 85 | 55.95 (68.44) | 46.51 (26.006) | 1090.10 (5491.94)
  Seq 2: Predose 0 hrs, Day 85: number analyzed (Participants) | 30 | 25 | 31
  Seq 2: Predose 0 hrs, Day 85 | 49.37 (52.93) | 1493.67 (4939.87) | 258.34 (1052.19)
  Seq 1+2: Predose 0 hrs, Day 85: number analyzed (Participants) | 61 | 53 | 60
  Seq 1+2: Predose 0 hrs, Day 85 | 52.72 (60.88) | 729.14 (3434.37) | 660.36 (3879.76)
  Seq 1: Postdose 0.08 Hrs, Day 29 and Day 57: number analyzed (Participants) | 34 | 35 | 31
  Seq 1: Postdose 0.08 Hrs, Day 29 and Day 57 | 42.51 (37.29) | 10967.36 (8543.58) | 22717.98 (16899.70)
  Seq 2: Postdose 0.08 Hrs, Day 29 and Day 57: number analyzed (Participants) | 31 | 24 | 33
  Seq 2: Postdose 0.08 Hrs, Day 29 and Day 57 | 278.61 (1278.26) | 16094.13 (12895.48) | 23107.50 (17012.10)
  Seq 1+2: Postdose 0.08 Hrs, Day 29 and Day 57: number analyzed (Participants) | 65 | 59 | 64
  Seq 1+2: Postdose 0.08 Hrs, Day 29 and Day 57 | 155.11 (883.60) | 13382.32 (10834.41) | 22918.34 (16823.84)
  Seq 1: Postdose 0.5 Hrs, Day 85: number analyzed (Participants) | 0 | 0 | 0
  Seq 2: Postdose 0.5 Hrs, Day 85: number analyzed (Participants) | 31 | 26 | 31
  Seq 2: Postdose 0.5 Hrs, Day 85 | 415.01 (1990.46) | 9508.98 (6547.42) | 26420.12 (16539.03)
  Seq 1+2: Postdose 0.5 Hrs, Day 85: number analyzed (Participants) | 31 | 26 | 31
  Seq 1+2: Postdose 0.5 Hrs, Day 85 | 415.01 (1990.46) | 9508.98 (6547.42) | 26420.12 (16539.03)
  Seq 1: Postdose 1 Hr, Day 1: number analyzed (Participants) | 35 | 38 | 33
  Seq 1: Postdose 1 Hr, Day 1 | 483.03 (2593.24) | 4761.62 (5209.23) | 14623.63 (13535.30)
  Seq 2: Postdose 1 Hr, Day 1: number analyzed (Participants) | 0 | 0 | 0
  Seq 1+2: Postdose 1 Hr, Day 1: number analyzed (Participants) | 35 | 38 | 33
  Seq 1+2: Postdose 1 Hr, Day 1 | 483.03 (2593.24) | 4761.62 (5209.23) | 14623.63 (13535.30)
  Seq 1: Postdose 1.5 Hrs, Day 29: number analyzed (Participants) | 0 | 0 | 0
  Seq 2: Postdose 1.5 Hrs, Day 29: number analyzed (Participants) | 33 | 29 | 32
  Seq 2: Postdose 1.5 Hrs, Day 29 | 27.28 (24.42) | 3086.34 (4433.97) | 6337.84 (5955.82)
  Seq 1+2: Postdose 1.5 Hrs, Day 29: number analyzed (Participants) | 33 | 29 | 32
  Seq 1+2: Postdose 1.5 Hrs, Day 29 | 27.28 (24.42) | 3086.34 (4433.97) | 6337.84 (5955.82)
  Seq 1: Postdose 3 Hrs, Day 85: number analyzed (Participants) | 30 | 30 | 27
  Seq 1: Postdose 3 Hrs, Day 85 | 43.80 (72.69) | 1137.22 (3218.04) | 2415.05 (5479.82)
  Seq 2: Postdose 3 Hrs, Day 85: number analyzed (Participants) | 0 | 0 | 0
  Seq 1+2: Postdose 3 Hrs, Day 85: number analyzed (Participants) | 30 | 30 | 27
  Seq 1+2: Postdose 3 Hrs, Day 85 | 43.80 (72.69) | 1137.22 (3218.04) | 2415.05 (5479.83)
  Seq 1: Postdose 4 Hrs, Day 1: number analyzed (Participants) | 0 | 0 | 0
  Seq 2: Postdose 4 Hrs, Day 1: number analyzed (Participants) | 34 | 33 | 38
  Seq 2: Postdose 4 Hrs, Day 1 | 52.99 (64.23) | 1156.16 (2859.47) | 473.67 (1038.69)
  Seq 1+2: Postdose 4 Hrs, Day 1: number analyzed (Participants) | 34 | 33 | 38
  Seq 1+2: Postdose 4 Hrs, Day 1 | 52.99 (64.23) | 1156.16 (2859.47) | 473.67 (1038.69)
  Seq 1: Postdose 6 Hrs, Day 57: number analyzed (Participants) | 32 | 31 | 29
  Seq 1: Postdose 6 Hrs, Day 57 | 51.39 (71.32) | 304.67 (1157.61) | 431.94 (1282.37)
  Seq 2: Postdose 6 Hrs, Day 57: number analyzed (Participants) | 0 | 0 | 0
  Seq 1+2: Postdose 6 Hrs, Day 57: number analyzed (Participants) | 32 | 31 | 29
  Seq 1+2: Postdose 6 Hrs, Day 57 | 51.39 (71.32) | 304.67 (1157.61) | 431.94 (1282.37)

8. Secondary Outcome: Absolute Concentrations of SUN11031 Metabolites Desacyl-ghrelin Following Treatment With SUN11031 in Participants Having Cachexia Associated With Chronic Obstructive Pulmonary Disease
Description: Absolute concentrations of SUN11031 metabolites desacyl-ghrelin in participant plasma samples were measured. When participants were randomly assigned into 1 of 3 treatment groups at baseline, they were also randomly assigned into 1 of 2 sequences in the pharmacokinetic (PK) sparse sampling schedule based on the randomization number.
Time Frame: as for outcome 7
Population: Absolute concentrations of SUN11031 metabolites were assessed using the pharmacokinetic population.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg
Number analyzed (Participants) | 73 | 74 | 76
pg/mL
  Seq 1: Predose 0 hrs, Day 1: number analyzed (Participants) | 36 | 36 | 29
  Seq 1: Predose 0 hrs, Day 1 | 189.79 (170.09) | 351.53 (1102.43) | 547.12 (1276.89)
  Seq 2: Predose 0 hrs, Day 1: number analyzed (Participants) | 34 | 32 | 37
  Seq 2: Predose 0 hrs, Day 1 | 175.88 (135.75) | 754.23 (3103.32) | 234.63 (225.77)
  Seq 1+2: Predose 0 hrs, Day 1: number analyzed (Participants) | 70 | 68 | 66
  Seq 1+2: Predose 0 hrs, Day 1 | 183.03 (153.42) | 541.04 (2265.36) | 371.94 (868.91)
  Seq 1: Predose 0 hrs, Day 85: number analyzed (Participants) | 31 | 29 | 29
  Seq 1: Predose 0 hrs, Day 85 | 207.81 (227.93) | 196.17 (131.67) | 951.98 (3846.40)
  Seq 2: Predose 0 hrs, Day 85: number analyzed (Participants) | 29 | 25 | 30
  Seq 2: Predose 0 hrs, Day 85 | 158.60 (131.94) | 459.03 (1059.43) | 824.12 (3095.66)
  Seq 1+2: Predose 0 hrs, Day 85: number analyzed (Participants) | 60 | 54 | 59
  Seq 1+2: Predose 0 hrs, Day 85 | 184.03 (187.86) | 317.86 (731.38) | 886.97 (3455.15)
  Seq 1: Postdose 0.08 Hrs, Day 29 and Day 57: number analyzed (Participants) | 32 | 35 | 31
  Seq 1: Postdose 0.08 Hrs, Day 29 and Day 57 | 174.87 (186.0) | 5401.49 (4793.51) | 8680.49 (7747.93)
  Seq 2: Postdose 0.08 Hrs, Day 29 and Day 57: number analyzed (Participants) | 32 | 25 | 32
  Seq 2: Postdose 0.08 Hrs, Day 29 and Day 57 | 292.21 (655.71) | 6560.23 (4751.75) | 9519.43 (8835.18)
  Seq 1+2: Postdose 0.08 Hrs, Day 29 and Day 57: number analyzed (Participants) | 64 | 60 | 63
  Seq 1+2: Postdose 0.08 Hrs, Day 29 and Day 57 | 233.54 (481.75) | 5884.30 (4770.54) | 9106.62 (8261.72)
  Seq 1: Postdose 0.5 Hrs, Day 85: number analyzed (Participants) | 0 | 0 | 0
  Seq 2: Postdose 0.5 Hrs, Day 85: number analyzed (Participants) | 30 | 26 | 31
  Seq 2: Postdose 0.5 Hrs, Day 85 | 417.51 (1407.84) | 6200.68 (5045.86) | 10819.65 (7950.18)
  Seq 1+2: Postdose 0.5 Hrs, Day 85: number analyzed (Participants) | 30 | 26 | 31
  Seq 1+2: Postdose 0.5 Hrs, Day 85 | 417.51 (1407.84) | 6200.68 (5045.86) | 10819.65 (7950.18)
  Seq 1: Postdose 1 Hr, Day 1: number analyzed (Participants) | 35 | 37 | 32
  Seq 1: Postdose 1 Hr, Day 1 | 438.24 (1658.63) | 3071.61 (2422.07) | 7929.87 (7053.81)
  Seq 2: Postdose 1 Hr, Day 1: number analyzed (Participants) | 0 | 0 | 0
  Seq 1+2: Postdose 1 Hr, Day 1: number analyzed (Participants) | 35 | 37 | 32
  Seq 1+2: Postdose 1 Hr, Day 1 | 438.24 (1658.63) | 3071.61 (2422.07) | 7929.87 (7053.81)
  Seq 1: Postdose 1.5 Hrs, Day 29: number analyzed (Participants) | 0 | 0 | 0
  Seq 2: Postdose 1.5 Hrs, Day 29: number analyzed (Participants) | 33 | 30 | 33
  Seq 2: Postdose 1.5 Hrs, Day 29 | 105.15 (77.91) | 2230.16 (1920.22) | 4944.39 (4285.93)
  Seq 1+2: Postdose 1.5 Hrs, Day 29: number analyzed (Participants) | 33 | 30 | 33
  Seq 1+2: Postdose 1.5 Hrs, Day 29 | 105.15 (77.91) | 2230.16 (1290.22) | 4944.39 (4285.93)
  Seq 1: Postdose 3 Hrs, Day 85: number analyzed (Participants) | 29 | 30 | 29
  Seq 1: Postdose 3 Hrs, Day 85 | 128.21 (147.42) | 2381.54 (4226.73) | 2536.51 (1949.44)
  Seq 2: Postdose 3 Hrs, Day 85: number analyzed (Participants) | 0 | 0 | 0
  Seq 1+2: Postdose 3 Hrs, Day 85: number analyzed (Participants) | 29 | 30 | 29
  Seq 1+2: Postdose 3 Hrs, Day 85 | 128.21 (147.42) | 2381.54 (4226.73) | 2536.51 (1949.44)
  Seq 1: Postdose 4 Hrs, Day 1: number analyzed (Participants) | 0 | 0 | 0
  Seq 2: Postdose 4 Hrs, Day 1: number analyzed (Participants) | 37 | 32 | 39
  Seq 2: Postdose 4 Hrs, Day 1 | 132.97 (126.11) | 1071.31 (1124.55) | 993.47 (1167.56)
  Seq 1+2: Postdose 4 Hrs, Day 1: number analyzed (Participants) | 37 | 32 | 39
  Seq 1+2: Postdose 4 Hrs, Day 1 | 132.97 (126.11) | 1071.31 (1124.55) | 993.47 (1167.56)
  Seq 1: Postdose 6 Hrs, Day 57: number analyzed (Participants) | 31 | 30 | 28
  Seq 1: Postdose 6 Hrs, Day 57 | 149.58 (166.07) | 577.37 (632.84) | 914.64 (769.17)
  Seq 2: Postdose 6 Hrs, Day 57: number analyzed (Participants) | 0 | 0 | 0
  Seq 1+2: Postdose 6 Hrs, Day 57: number analyzed (Participants) | 31 | 30 | 28
  Seq 1+2: Postdose 6 Hrs, Day 57 | 149.58 (166.07) | 577.37 (632.84) | 914.64 (769.17)

9. Secondary Outcome: Treatment Emergent Adverse Events Reported in ≥ 2% of Participants Following Treatment With SUN11031 in Participants Having Cachexia Associated With Chronic Obstructive Pulmonary Disease
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that occurred from the time treatment was administered at Day 1 through the last follow-up visit or a worsening of a pre-existing condition.
Time Frame: Baseline up to Day 113 post dose, up to a total of 134 days.
Population: Treatment-emergent adverse events were assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg
Number analyzed (Participants) | 73 | 75 | 76
Participants
  Number of Participants with at least 1 TEAE | 58 | 59 | 56
  COPD | 23 | 20 | 16
  Dyspnea | 1 | 2 | 3
  Bronchitis | 4 | 5 | 3
  Nasopharyngitis | 1 | 6 | 2
  Influenza | 2 | 3 | 3
  Pneumonia | 1 | 2 | 3
  Gastroenteritis | 2 | 2 | 2
  Urinary tract infection | 2 | 1 | 3
  upper respiratory tract infection | 3 | 1 | 2
  Pharyngitis | 1 | 0 | 2
  Sinusitis | 2 | 1 | 0
  Tonsillitis | 2 | 1 | 0
  Oral herpes | 2 | 0 | 0
  Diarrhea | 7 | 2 | 1
  Nausea | 3 | 1 | 5
  Abdominal pain upper | 0 | 4 | 3
  Toothache | 2 | 0 | 2
  Abdominal pain | 1 | 2 | 0
  Dry mouth | 1 | 0 | 2
  Vomiting | 2 | 0 | 1
  Injection site hematoma | 7 | 3 | 7
  Injection site pain | 2 | 4 | 2
  Chest pain | 1 | 2 | 1
  Asthenia | 3 | 0 | 1
  Thirst | 0 | 0 | 2
  Back pain | 1 | 4 | 3
  Arthralgia | 1 | 1 | 2
  Myalgia | 2 | 2 | 0
  Muscle spasms | 0 | 1 | 2
  Hepatic enzyme increased | 1 | 2 | 0
  Weight decreased | 3 | 6 | 4
  Electrocardiogram QT prolonged | 2 | 0 | 1
  Headache | 5 | 4 | 5
  Dizziness | 1 | 2 | 3
  Hypertension | 4 | 1 | 1
  Hypotension | 2 | 1 | 1
  Orthostatic hypotension | 0 | 2 | 0
  Sinus tachycardia | 0 | 2 | 0
  Hyperglycemia | 2 | 2 | 1
  Hyperkalemia | 1 | 2 | 0
  Insomnia | 1 | 0 | 4
  Somnolence | 2 | 0 | 1
  Depression | 0 | 0 | 2
  Hyperhidrosis | 0 | 2 | 4
  Contusion | 0 | 0 | 2
  Cholecystitis | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline up to Day 113 post dose, up to a total of 134 days.
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that occurred from the time treatment was administered at Day 1 through the last follow-up visit or a worsening of a pre-existing condition.
Arm/Group | Placebo | SUN11031 20 μg/kg | SUN11031 40 μg/kg
All-Cause Mortality (participants affected / at risk) | 1/73 | 0/75 | 2/76
Serious Adverse Events (participants affected / at risk) | 6/73 | 6/75 | 8/76
Other Adverse Events (participants affected / at risk) | 54/73 | 54/75 | 47/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | SUN11031 20 μg/kg (N=75) | SUN11031 40 μg/kg (N=76)
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
COPD (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Senile dementia (Nervous system disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | SUN11031 20 μg/kg (N=75) | SUN11031 40 μg/kg (N=76)
COPD (Respiratory, thoracic and mediastinal disorders) | 23 | 20 | 16
Injection site hematoma (Injury, poisoning and procedural complications) | 7 | 3 | 7
Headache (Nervous system disorders) | 5 | 4 | 5
Weight decreased (Investigations) | 3 | 6 | 4
Bronchitis (Infections and infestations) | 4 | 5 | 3
Diarrhea (Gastrointestinal disorders) | 7 | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 6 | 2
Nausea (Gastrointestinal disorders) | 3 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3
Injection site pain (General disorders) | 2 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4 | 3
Hypertension (Vascular disorders) | 4 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No